CLINICAL TRIAL: NCT02742155
Title: Play2Sleep: A Sequential Explanatory Mixed Methods Study of Using Infant Play to Improve Infant Sleep in Families Experiencing Infant Sleep Disturbance
Brief Title: Play2Sleep: Using Play to Improve Infant Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Karen Benzies, Dr., University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB15-2652
Record Dates: First submitted 2016-04-05; First posted 2016-04-18 (Estimated); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Disturbances in Initiating and Maintaining Sleep; Parent-Child Relations
Keywords: Family Research

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Play2Sleep (Experimental): For the experimental intervention, Play2Sleep consists of video-recording the mother and father separately while engaged in a structured play session. Immediately following the play session, the home visitor will review the video recording with each parent separately to provide positive feedback on parental behaviors that promotes contingent interaction and identification of infant cues. At the end of the visit, standard public health handouts on infant sleep will be provided to both parents.
  Interventions: Behavioral: Play2Sleep
- Comparison (Active Comparator): In the comparison group, only standard public health handouts on infant sleep will be reviewed with parents.
  Interventions: Behavioral: Comparison

INTERVENTIONS:
Behavioral: Play2Sleep — Behavioral: Video self-modelling
  Arms: Play2Sleep
Behavioral: Comparison — Behavioral: Information only
  Arms: Comparison

SUMMARY:
The objective of this study is to evaluate and explore the effectiveness of Play2Sleep on families of infants with infant sleep disturbances.

DETAILED DESCRIPTION:
RESEARCH OBJECTIVE AND QUESTIONS:

The objective of this study is to evaluate and explore the effectiveness of Play2Sleep on families of infants with infant sleep disturbances.

The quantitative research question is: Does one dose of Play2Sleep delivered during home visits with mothers and fathers of 5-month-old infants with infant sleep disturbances reduce the number of night wakings at age 7 months? The qualitative phase will focus on explaining the quantitative findings by asking: What are parental perceptions of family experiences, processes, and contexts related to Play2Sleep and infant sleep? The overarching mixed methods research question is: How do parental perceptions of family experiences, processes, and contexts related to infant sleep explain the effectiveness of Play2Sleep?

METHODS:

An explanatory sequential mixed methods design will be used. The quantitative phase will be a pilot randomized controlled trial and the subsequent qualitative phase will employ Thematic Analysis of parental interviews to understand their perspectives on the effectiveness and acceptability of Play2Sleep.

Public health nurses will introduce potential participants to the study during 4-month well-baby clinic visits. Inclusion criteria will be English-speaking mothers and fathers of healthy infants who perceive that their child has sleep problems. A total of 60 mother-father-infant triads with complete data will be obtained: 30 intervention; 30 comparison.

The experimental intervention, Play2Sleep, will occur during a home visit when the infant is 5 months old and will consist of video-recording each parent engaging in a structured play session with their infant. Immediately following the interaction sequence, the video-recording will be reviewed with the parent. Positive feedback on parental behaviors that promote interaction and child development will be provided during the video review. This will include the identification of the infant's social and sleep related cues. In addition to the standard public health handout on infant sleep, a handout on parent-infant behaviours will be given to encourage one or two areas that parents can continue to develop. During the video-recording and review, the other parent will not be present. The structured play sequence will follow established protocols in the Parent-Child Interaction Teaching Scale manual. The comparison group will receive only the standard public health handout.

Based on maximum and minimum changes in infant sleep, 20 families (10 intervention families and 10 comparison families) will be invited to participate in evaluative qualitative interviews upon completing the second home visit. Semi-structured family interviews will elicit descriptions about parental experiences that explain the quantitative findings. Interview will be transcribed and transcripts will be analyzed using Thematic Analysis. Preliminary results of the thematic analysis will be submitted to the qualitative participants for review and opportunities for clarification or further explication will be provided.

The quantitative and qualitative results will then be integrated together to draw overarching conclusions about the effectiveness of Play2Sleep. Specifically, the results from the qualitative interviews will be used to explain and contextualize the quantitative results.

ELIGIBILITY:
Inclusion Criteria:

* co-habiting mothers and fathers of full-term, healthy, singleton, 4-month old infants
* first-time parents
* able to read, write, and speak English
* perceive that their infant has sleep disturbances
* whose infant experiences one of the following: (a) greater than 3 night wakings per night; (b) awake greater than 60 minutes during the night; or (c) less than 9 hours total day and night time sleep.

Exclusion Criteria:

* a known or suspected medical or physiological cause of sleep problems in either parent or infant

Ages: 4 Months to 5 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 136 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-07-23 (Actual); Study Completion 2018-07-23 (Actual)

PRIMARY OUTCOMES:
Infant night wakings using the Brief Infant Sleep Questionnaire | 2 months
  As provided by parental report using the Expanded version of the Brief Infant Sleep Questionnaire

SECONDARY OUTCOMES:
Parental report of infant sleep patterns using the Brief Infant Sleep Questionnaire | 2 months
  As provided by parental report using the Expanded version of the Brief Infant Sleep Questionnaire.
Parental depression using the Edinburgh Postnatal Depression Scale (EPDS) | 2 months
Parental Sense of Competence using the Parental Sense of Competence (PSOC) Scale | 2 months
Marital satisfaction using the brief version of the Dyadic Adjustment Scale (DAS-4) | 2 months
Parent-child interactions using the Parent-Child Interaction Teaching Scale (PCITS) | 2 months
  The PCITS is a 73-item coding scheme of a structured parent-child play session that measure the quality of parent-child interactions. Play sessions follow established protocols in the Parent-child interaction teaching scale manual and are video recorded for later coded according to the PCITS items. The PCITS includes 4 parent sub-scales (sensitivity, response to child's distress, social-emotional growth fostering, and cognitive growth fostering) and 2 child sub-scales (clarity of cues and responsiveness to caregiver).
Parental cognitions about infant sleep using the Maternal Cognitions about Infant Sleep Questionnaire (MCISQ) | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Karen M Benzies, PhD, Principal Investigator — University of Calgary
Locations (9):
- Canada (9):
  - Village Square Community Health Centre, Calgary, Alberta
  - East Calgary Health Centre, Calgary, Alberta
  - Acadia Community Health Centre, Calgary, Alberta
  - Thornhill Community Health Centre, Calgary, Alberta
  - University of Calgary, Calgary, Alberta
  - Sheldon M. Chumir Health Centre, Calgary, Alberta
  - South Calgary Health Centre, Calgary, Alberta
  - Shaganappi Community Health Centre, Calgary, Alberta
  - Northwest Community Health Centre, Calgary, Alberta

IPD SHARING:
Plan to Share IPD: Yes
Following study completion, de-identified data will be submitted to SAGE at Policy Wise (formerly the Child Data Centre of Alberta), a research and data facility operating under the authority of the Alberta Centre for Child, Family and Community Research.

REFERENCES:
- [Derived] Keys EM, Benzies KM, Kirk VG, Duffett-Leger L. Effect of Play2Sleep on mother-reported and father-reported infant sleep: a sequential explanatory mixed-methods study of a randomized controlled trial. J Clin Sleep Med. 2022 Feb 1;18(2):439-452. doi: 10.5664/jcsm.9618. PMID 34409935
- [Derived] Keys E, Benzies KM, Kirk V, Duffett-Leger L. Using Play to Improve Infant Sleep: A Mixed Methods Protocol to Evaluate the Effectiveness of the Play2Sleep Intervention. Front Psychiatry. 2018 Apr 17;9:109. doi: 10.3389/fpsyt.2018.00109. eCollection 2018. PMID 29719517